CLINICAL TRIAL: NCT05636709
Title: National Post-market Clinical Follow-up Study to Evaluate in Real-world Practice the Efficacy and Safety of Granulocytoapheresis and Its Impact on Quality of Life in Patients With Inflammatory Bowel Disease
Brief Title: National GMA Post-market Clinical Follow-up Study (GRACE)
Acronym: GRACE
Status: Recruiting | Type: Observational
Sponsor: Adacyte Therapeutics SL (Industry)
Responsible Party: Sponsor
Other Study IDs: GRACE
Record Dates: First submitted 2022-08-24; First posted 2022-12-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Adacolumn — Non interventional study

SUMMARY:
Inflammatory bowel disease (IBD) encompasses several chronic diseases of which ulcerative colitis (UC) and Crohn's disease (CD) are the most representative. IBD is characterised by the presence of an inflammatory process that affects different segments of the digestive tract and has a chronic and relapsing course with flares of activity.

Inflammatory activity in IBD is associated with an increase in peripheral blood activated granulocytes and monocyte-macrophages and intestinal infiltration by these inflammatory cells, which are largely responsible for tissue damage. In recent years, observational, prospective studies and meta-analyses of these studies have contributed to consider granulocytapheresis (GMA) as an effective and safe alternative in the treatment of UC.

This apheresis technique is based on recirculation of the patient's blood through a circuit with cellulose acetate spheres that perform a selective elimination of granulocytes and monocyte-macrophages leading to a reduction in pro-inflammatory cytokines and adhesion molecule expression, and an increase in anti-inflammatory mediators. These events in the GMA column are followed by other immunological changes, most notably a decrease in CD10+ (activated) neutrophils, leading to a compensation from the bone marrow of a CD10- (immature) neutrophil population.

GMA can be considered as a therapeutic alternative in corticodependent IBD, especially in UC. In addition, it can reduce or limit the need for corticosteroids, so another possible application is as a "bridge" treatment in patients starting treatment with thiopurine immunomodulators. A beneficial effect can also be obtained by combining apheresis with biological treatments, especially after a partial response or loss of response to these treatments. Finally, some extraintestinal manifestations associated with IBD may also benefit from its use.

The GRACE study is proposed for the evaluation of the efficacy of GMA with Adacolumn® under real conditions of use and according to the indications described in the instructions for use of the medical device.

DETAILED DESCRIPTION:
It is planned to enrol a minimum of 350 patients from approximately 30 sites. To avoid screening biases, the patients to be included per site will be selected consecutively from among those who meet the eligibility criteria to participate in the study.

A national, multicentre, noninterventional post-market clinical follow-up (PMCF) study with an estimated follow-up period of 12 months after completion of GMA therapy to evaluate the efficacy of Adacolumn® GMA in actual conditions of use, as specified in the product instructions for use, in adult patients diagnosed with UC or CD. Approximately 350 patients from about 30 centres in Spain are planned to be included.

The standard regimen according to product instructions for use is one session per week for 5 consecutive weeks, although in specific cases continuous regimens have been established for maintenance (one or two sessions per month) or others for induction (two sessions per week). The use of a higher number of sessions seems to increase efficacy from 40% with 5 sessions to 80% with 10 in the more refractory cases and may achieve a greater reduction in steroid use. In Europe, where GMA is used in different scenarios, it is routinely being used in 7 to 10 sessions.

The study will consist of a maximum of 4 visits: a baseline visit, which will coincide with patient inclusion in the study, and 3 follow-up visits at 4 (±2 weeks) (month 1), 24 (±2 weeks) (month 6) and 48 (±2 weeks) (month 12) weeks after the last session of induction apheresis.

All visits scheduled during the study will coincide with any of the patient visits made as part of routine clinical follow-up, without interfering with the investigator's clinical duties. Note: In the event that a patient discontinues Adacolumn® GMA, the reasons for discontinuation of the procedure will be recorded and the change in treatment for IBD, if any.

Once the patient has been adequately informed, his/her eligibility has been confirmed and he/she has signed the informed consent (IC), the investigator will start data collection in an appropriate and precise manner. Therefore, no diagnostic or therapeutic intervention outside of routine clinical practice will be applied. To ensure the noninterventional nature of the study, the data will be collected provided they are available in the patient's medical record or can be collected during patient visits to his/her physician as part of actual clinical care (as in the case of questionnaires used as source documents).

Adacolumn® is a medical device intended for modifying the biological or chemical composition of the blood (class IIb), according to Regulation (UE) 2017/745 on Medical Devices, manufactured by Japan Immnunoresearch Laboratories, JIMRO (Takasaki, Japan). It consists of a 335 ml column formed by cellulose acetate beads of 2 mm in diameter bathed in saline, where granulocytes (65%), monocytes (55%), and only 2% of lymphocytes are selectively adsorbed.

Adacolumn® is indicated for induction of remission in patients with IBD (active UC and CD), for suppression of subjective and objective symptoms in patients with rheumatoid arthritis in the inflammatory stage whose symptoms might be resistant to standard drug therapy, for treatment of patients with ocular Behcet disease and for treatment of patients with systemic lupus erythematosus.

In this study, the intended use of Adacolumn® is for application of GMA in patients diagnosed with IBD, both UC and CD

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years.
2. Established diagnosis of UC or CD according to ECCO criteria.
3. Patients in whom the physician in charge of treatment decides to start treatment with GMA and independently of their inclusion in the study.
4. Patients who understand and voluntarily sign informed consent.

Exclusion Criteria:

1. Patient with any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to comply with the study procedures.
2. Patient who is participating in a clinical trial.

NOTE: If the physician knows or suspects that the patient is unable to understand the implications of his/her participation in the study, the patient should not enter without the signature of his/her legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Ulcerosis Colitis or Crohn disease from about 30 centres in Spain in whom the physician in charge of treatment decides to start treatment with GMA and independently of their inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving steroid-free clinical remission at 6 months after completion of GMA therapy | 6 months
  Proportion of patients achieving steroid-free clinical remission at 6 months after completion of GMA therapy. Clinical remission is defined as:
  1. For Ulcerative Colitis: Total Mayo score ≤2, with no subscore >1 and rectal bleeding subscore of 0.
  2. For Crohn´s Disease: Harvey-Bradshaw Index score ≤4.
  Mayor score (0-12). Higher scores mean a worse outcome. Harvey-Bradshaw Index (0-undetermined). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Define the regimens used for GMA in actual clinical practice. | 12 months
  The strategies for use of GMA will be evaluated by the following:
  * Frequency of GMA sessions, Number of sessions, Blood volume processed per session in ml, Length of sessions in minutes, Method of administration of the technique (peripheral access or central catheter), Type of anticoagulant (Heparin, sodic heparin, low molecular weight heparin), Dose of anticoagulant (ml), Form of administration (infusion or bolus).
  * Proportion of patients receiving GMA treatment combined with biologics or immunosuppressants as bridge treatment after instituting treatment with immunomodulators due to lack of response or intolerance to immunosuppressants and/or biologics or as an alternative to conventional treatment.
  * Proportion of patients with steroid-dependent or steroid-refractory disease receiving GMA.
  * Proportion of patients receiving GMA as treatment for remission induction or relapse prevention.
  * Proportion of patients receiving GMA as maintenance treatment
Early clinical remission rate | 1 month
  Proportion of patients achieving steroid-free clinical remission at 1 month after completion of GMA therapy
  Clinical remission is defined as:
  1. For Ulcerative Colitis: Total Mayo score ≤2, with no subscore >1 and rectal bleeding subscore of 0.
  2. For Crohn´s Disease: Harvey-Bradshaw Index score ≤4.
  Mayor score (0-12). Higher scores mean a worse outcome. Harvey-Bradshaw Index (0-undetermined). Higher scores mean a worse outcome.
6- and 12-month remission rates completion of GMA therapy | 6 and 12-month
  Proportion of patients achieving steroid-free clinical remission at 12 months after completion of GMA therapy
  Clinical remission is defined as:
  1. For Ulcerative Colitis: Total Mayo score ≤2, with no subscore >1 and rectal bleeding subscore of 0.
  2. For Crohn´s Disease: Harvey-Bradshaw Index score ≤4.
  Mayor score (0-12). Higher scores mean a worse outcome. Harvey-Bradshaw Index (0-undetermined). Higher scores mean a worse outcome.
Sustained clinical remission rate | 12 months
  Proportion of patients maintaining clinical remission at 12 months after completion of GMA therapy
  Clinical remission at 12 months is defined as:
  1. For Ulcerative Colitis: Total Mayo score ≤2, with no subscore >1 and rectal bleeding subscore of 0.
  2. For Crohn´s Disease: Harvey-Bradshaw Index score ≤4.
  Until 12 months
  Mayor score (0-12). Higher scores mean a worse outcome. Harvey-Bradshaw Index (0-undetermined). Higher scores mean a worse outcome.
6- and 12-month clinical response rates | 6 and 12-month
  Proportion of patients with clinical response at 6 and 12 months after completion of GMA therapy, defined as a reduction of 3 o more points or 30% in the Mayo score for Ulcerative Colitis, or 3 or more points in the Harvey Bradshaw index for Crohn´s Disease
  Mayor score (0-12) Harvey-Bradshaw Index (0-undetermined) Higher scores mean a worse outcome.
Rate of patients receiving GMA as maintenance and its efficacy | 12 months
  Proportion of patients on maintenance treatment remaining in steroid-free clinical remission at 6 (visit 3) and 12 (visit 4) months after completion of therapy
  Clinical remission is defined as:
  1. For Ulcerative Colitis: Total Mayo score ≤2, with no subscore >1 and rectal bleeding subscore of 0.
  2. For Crohn´s Disease: Harvey-Bradshaw Index score ≤4.
  At 6 months and 12 months Mayor score (0-12). Higher scores mean a worse outcome. Harvey-Bradshaw Index (0-undetermined). Higher scores mean a worse outcome.
Rate of patients requiring steroids and mean dose during follow-up | 12 months
  * Rate of patients requiring steroids
  * Mean dose of steroids
  Steroids in mg
Changes in faecal calprotectin and C-reactive protein (CRP) biomarkers during treatment | 12 months
  The change in biomarkers levels (faecal calprotectin (microg/g or mg/Kg) and CRP (mg/L)) will be evaluated by laboratory tests performed at the baseline visit (visit 1), at each apheresis session, at 1 month after completion of treatment (visit 2) and at 6 (visit 3) and 12 months (visit 4) after completion of treatment.
Rate of treatment-related adverse events (AEs) and seriousness | 6 months
  Frequency of treatment-related AEs and seriousness
Change in patients' quality of life | 6 months
  The change in quality of life will be evaluated by the validated version in Spanish of the Inflammatory Bowel Disease Questionnaire, which will be completed by the patient at the baseline visit (visit 1), at each apheresis session, at 1, (visit 2), 6 (visit 3) and 12 months (visit 4) after completion of treatment
  Inflammatory Bowel Disease Questionnaire (0-100) Higher scores mean a better outcome.
Number of patients requiring surgery | 6 months
  Proportion of patients requiring surgery during the study period (UC: colectomy, segmental colonic resection, perianal; CD: small intestine resection, colonic resection, ileocecal resection, perianal resection).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Cabriada, Study Chair — H. Galdakao; Iago Rodríguez, Study Chair — H. Galdakao; Daniel Ginard, Study Chair — H. Son Espases
Locations (30):
- Spain (30):
  - H. Albacete, Albacete, Albacete
  - H. General de Alicante, Alicante, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - H. Vall d´hebron, Barcelona, Barcelona
  - H. Galdakao, Galdakao, Bizkaia
  - H. General de Castellón, Castellon, Castellón
  - H. Puerta del Mar, Cadiz, Cádiz
  - H. Reina Sofía, Córdoba, Córdoba
  - H. Donostia, San Sebastián, Gipuzkoa
  - H. Virgen de las Nieves, Granada, Granada
  - H. Guadalajara, Guadalajara, Guadalajara
  - H. San Jorge, Huesca, Huesca
  - H. Santiago, Santiago de Compostela, La Coruña
  - H. San Pedro, Logroño, La Rioja
  - H. Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas de Gran Canarias
  - H. 12 de octubre, Madrid, Madrid
  - H. La Paz, Madrid, Madrid
  - H. Costa del Sol, Marbella, Málaga
  - H. Navarra, Pamplona, Navarre
  - H. Río Carrión, Palencia, Palencia
  - H. Son Espases, Palma de Mallorca, Palma de Mallorca
  - H. Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - H. Álvaro Cunqueiro, Vigo, Pontevedra
  - H. Univ. de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - H. Ntra. Sra. de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - H. Virgen del Rocío, Seville, Sevilla
  - H. Clínico Univ. de Valencia, Valencia, Valencia
  - H. General de Valencia, Valencia, Valencia
  - H. La Fe, Valencia, Valencia
  - H. Virgen de la Concha, Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No